CLINICAL TRIAL: NCT04770935
Title: A Phase 1, Open-Label Study to Assess the Pharmacokinetics, and Safety and Tolerability of a Single Intravenous Injection of rFVIIIFc-VWF-XTEN (BIVV001) in Adults With Type 2N and 3 Von Willebrand Disease (VWD)
Brief Title: To Assess the Pharmacokinetics and Safety and Tolerability of Efanesoctocog Alfa (BIVV001)in Adults With Type 2N and 3 Von Willebrand Disease (VWD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PKM16978; 2020-004947-10 (EudraCT Number); U1111-1255-4463 (Other: UTN)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Von Willebrand's Disease (VWD)
MeSH Terms: conditions — von Willebrand Diseases | interventions — BIVV001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- efanesoctocog alfa (BIVV001) (Experimental): A single IV dose of BIVV001 will be administered to each patient
  Interventions: Drug: efanesoctocog alfa (BIVV001)

INTERVENTIONS:
Drug: efanesoctocog alfa (BIVV001) — Pharmaceutical form:solution for injection Route of administration: intravenous injection

SUMMARY:
Primary Objective:

-To characterize the pharmacokinetics (PK) of BIVV001 after a single intravenous (IV) administration, as assessed by factor VIII (FVIII) activity determined by the one-stage activated partial thromboplastin time (aPPT) clotting assay, as well as, BIVV001 capture chromogenic Coatest FVIII activity assay

Secondary Objective:

-To assess the safety and tolerability of a single IV dose of BIVV001 in adult patients with type 2N and 3 VWD

DETAILED DESCRIPTION:
Duration of each part of the study for one participant:

Total study duration: Up to 57 days.

* Screening: up to 28 days.
* Up to 29 days of safety observation following the IV BIVV001 dose administration (this period includes PK sampling up to the first 10 days following administration).

ELIGIBILITY:
Inclusion criteria :

-- Male and/or female participant, between 18 and 65 years of age, inclusive at the time of informed consent.

* The participant has been diagnosed with hereditary type 3 VWD or type 2N VWD as documented in historical medical records OR a documented genotype known to produce VWD type 3 or 2N VWD.
* Type 3 VWD participants are included if they have a medical history of at least 25 exposure days to VWF and factor VIII-containing coagulation factor concentrates
* Type 2N VWD participants are included if the use of DDAVP is deemed insufficient or contraindicated, as assessed by the Investigator, or if they have required prior use of VWF- and FVIII- containing coagulation factor concentrates.

Exclusion criteria:

* Hereditary or acquired coagulation disorder other than VWD (including qualitative and quantitative platelet disorders, and thrombocytopenia < 100,000 cells/uL at Screening)
* The participant has a FVIII activity levels >20 IU/dL, at Screening
* History or presence of a VWF inhibitor or clinical suspicion of a VWF inhibitor
* History of a positive FVIII inhibitor test, defined as ≥0.6 BU/mL (by Nijmegen modified Bethesda assay) or a clinical suspicion of a FVIII inhibitor
* Positive FVIII inhibitor test, defined as ≥0.6 BU/mL, at Screening
* History of hypersensitivity or anaphylaxis associated with any FVIII- or VWF- containing product
* The participant has received or anticipates receiving systemic immunosuppressive or immunomodulatory treatment within 12 weeks prior to Baseline.
* The participant requires the use of acetylsalicylic acid, non-NSAID anti-platelets, and NSAIDs above the maximum dose product
* Patients currently on a prophylaxis regimen for the treatment of VWD that, in the Investigator's opinion, would preclude participation in the study due to the possible increased risk of bleeding associated with the requirement to withhold prophylaxis during the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Maximum plasma concentration observed (Cmax) | Day 1 to Day 10
Pharmacokinetic Parameter: Terminal half-life (t½z) | Day 1 to Day 10
Pharmacokinetic Parameter: Total Clearance (CL) | Day 1 to Day 10
Pharmacokinetic Parameter: Volume of distribution at steady state (Vss) | Day 1 to Day 10
Pharmacokinetic Parameter: Area under the activity time curve extrapolated to infinity (AUC∞) | Day 1 to Day 10
Pharmacokinetic Parameter: Mean residence time (MRT) | Day 1 to Day 10
Pharmacokinetic Parameter: Incremental recovery (IR) | Day 1 to Day 10

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (2):
  - University of Iowa_Investigational Site Number :8400002, Iowa City, Iowa
  - Hemophilia Center of Western Pennsylvania_Investigational Site Number :8400001, Pittsburgh, Pennsylvania
- France (2):
  - Investigational Site Number :2500001, Lille
  - Investigational Site Number :2500002, Nantes

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM16978 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25323&tenant=MT_SNY_9011